CLINICAL TRIAL: NCT06248411
Title: A Phase 1, Uncontrolled, Open-label, Non-randomized, Dose-escalation Study of KK2260 in Patients With Advanced or Metastatic Solid Tumors, Followed by an Uncontrolled, Non-randomized Study and an Uncontrolled, Randomized Study in Patients With Esophageal Squamous Cell Carcinoma or Head and Neck Squamous Cell Carcinoma
Brief Title: A Clinical Study of KK2260 in Patients With Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2260-001
Record Dates: First submitted 2023-09-26; First posted 2024-02-08 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Advanced or Metastatic Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KK2260 (Dosing regimen 1) (Experimental)
  Interventions: Drug: KK2260
- KK2260 (Dosing regimen 2) (Experimental)
  Interventions: Drug: KK2260

INTERVENTIONS:
Drug: KK2260 — KK2260 will be administered intravenously at several dose levels, and after determining MTD, multiple dose regimens will be evaluated in multiple cancer types to target.
  Arms: KK2260 (Dosing regimen 1)
Drug: KK2260 — KK2260 will be administered intravenously at several dose levels, and after determining MTD, multiple dose regimens will be evaluated in multiple cancer types to target.
  Arms: KK2260 (Dosing regimen 2)

SUMMARY:
This is the first in human study of KK2260. In Part 1a, the maximum tolerated dose (MTD) will be determined while evaluating the safety and tolerability of KK2260 in patients with advanced or metastatic solid tumors (any cancer type). In Part 1b and Part 2, at least three dosing regimens and two dosing regimens by cancer type, respectively, will be selected, and the safety, tolerability, and efficacy of each regimen will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

<Common Inclusion Criteria for Part 1a, Part 1b, and Part 2

1. Patients who have given informed written consent.
2. Male or female subjects ≥18 years of age, at time of signing informed consent.
3. Subjects who are refractory to standard treatment, intolerant of standard treatment, for whom standard treatment does not exist, or who have refused standard treatment.
4. Patients with measurable disease according to RECIST version 1.1
5. Patients who have had the certaion periods between the date of completion of prior therapy and the date of enrollment
6. Subjects who agree to have a tumor biopsy as part of the baseline examination. Patients who have difficulty in performing a tumour biopsy and have agreed to submit a previously collected stored specimen.
7. Patients with an ECOG PS of 0 or 1 at baseline.
8. Patients with haematopoietic, hepatic, renal, cardiac and respiratory functions that meet certain criteria in a baseline test.

<Additional Inclusion Criteria for Part 1a

1) Patients with pathologically diagnosed advanced or metastatic solid tumors.

<Additional Inclusion Criteria for Part 1b

1. Patients with pathologically diagnosed with advanced or metastatic esophageal cancer, or advanced or metastatic head and neck cancer whose primary site of origin is the oral cavity, oropharynx, hypopharynx, larynx, nasal cavity, or paranasal sinuses.
2. Patients with pathologically diagnosed squamous cell carcinoma.
3. Patients who agree to undergo tumor biopsy after administration.

<Additional Inclusion Criteria for Part 2a

1. Patients with pathologically diagnosed with advanced or metastatic esophageal cancer.
2. Patients with pathologically diagnosed squamous cell carcinoma.
3. Patients who agree to undergo tumor biopsy after administration.

<Additional Inclusion Criteria for Part 2b

1. Patients with advanced or metastatic head and neck cancer whose primary site of origin is the oral cavity, oropharynx, hypopharynx, larynx, nasal cavity, or paranasal sinuses.
2. Patients with pathologically diagnosed squamous cell carcinoma.
3. Patients who agree to undergo tumor biopsy after administration.

Exclusion Criteria:

<Common Exclusion Criteria to Part 1 and Part 2>

1. Patients with central or brain pia mater metastases that are untreated and symptomatic or that require treatment.
2. Patients with concurrent multiple or synchronous cancers, or with iatrogenic multiple or synchronous cancers with a disease-free interval of 5 years or less.
3. Patients receiving continuous systemic administration of steroids or other immunosuppressive drugs.
4. Patients who have had a Grade 3 or higher allergic reaction to an antibody agent or an additive of the study drug.
5. Patients who have not recovered to Grade 1 or below from adverse events caused by previously administered anticancer therapy.
6. Patients with active interstitial lung disease or a history of active interstitial lung disease.
7. Patients with infectious diseases requiring systemic treatment.
8. Patients with a fever of 38.0°C or higher at the time of registration.
9. Patients who test positive for Hepatitis B virus antigen or antibody, Hepatitis C virus antibody, or HIV antibody in a baseline test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2029-10-31 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (Only in Part 1a) | During the first cycle (1 Cycle = 28 days)
Adverse Events | Through study completion, an average of 1 year
Changes in Laboratory Testing Values (Red blood cell count) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Hemoglobin concentration) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Hematocrit) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Reticulocyte) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Mean corpuscular volume) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Mean corpuscular hemoglobin) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Mean corpuscular hemoglobin concentration) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (White blood cell count) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Differential white blood cells (basophils, eosinophils, lymphocytes, monocytes, neutrophils)) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Platelet count) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Total protein) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Albumin) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Alkaline phosphatase) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Alanine aminotransferase/Aspartate aminotransferase) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Total bilirubin/Direct bilirubin) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Blood urea nitrogen) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Calcium/Corrected Calcium) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Chloride) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Potassium) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Sodium) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Magnesium) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Serum iron) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Ferritin) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Total iron binding capacity) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Unsaturated iron binding capacity) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Serum creatinine) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Creatinine clearance (Cockgroft-gault formula)) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Lactate dehydrogenase) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Blood glucose) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Uric acid) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Lipase) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Amylase) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (C-reactive protein) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Gamma-glutamyl transpeptidase) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Triglycerides) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Cholesterol) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Creatine phosphokinase) | Every week through study completion, an average of 1 year
Changes in Laboratory Testing Values (Coagulation test) | Every week through study completion, an average of 1 year
  Prothrombin time international normalized ratio and Activated partial thromboplastin time
Changes in Laboratory Testing Values (Hepatitis B virus DNA, if needed) | Every 2 cycle through study completion, an average of 1 year (1 Cycle = 28 days)
Changes in Body temperature (degree Celsius) | Every week through study completion, an average of 1 year
Changes in Systolic and Diastolic Blood Pressure (mmHg) | Every week through study completion, an average of 1 year
Changes in SpO2 (%) | Every week through study completion, an average of 1 year
Changes in Electrocardiogram parameters (Heart rate, PR interval, QRS interval, QT interval, and QTc intervals) | Every week through study completion, an average of 1 year
  The resting Heart rate, PR interval, QRS interval, QT interval, and QTc intervals will be recorded. Any abnormalities in ECG will be specified and documented as clinically significant or not clinically significant.
Changes in Eastern Cooperative Oncology Group Performance Status (ECOG PS) (The score should be 0 to 4, and the lower is the better.) | Every week through study completion, an average of 1 year

SECONDARY OUTCOMES:
Serum concentration levels of KK2260 | Pre-dose and post-dose at multiple timepoints for each cycle during the intervention (each cycle is 28 days)
Maximum Plasma Concentration (Cmax) | Pre-dose and post-dose at multiple timepoints for each cycle during the intervention (each cycle is 28 days)
Area Under the blood concentration-time Curve (AUC) | Pre-dose and post-dose at multiple timepoints for each cycle during the intervention (each cycle is 28 days)
Anti-drug antibody | Pre-dose and post-dose at multiple timepoints for each cycle during the intervention (each cycle is 28 days)
Overall Response Rate (in Part 1b/2) | During the treatment and every 12 weeks after study treatment completion (approximately up to 1 year)
Disease Control Rate (in Part 1b/2) | During the treatment and every 12 weeks after study treatment completion (approximately up to 1 year)
Duration of Response (in Part 1b/2) | During the treatment and every 12 weeks after study treatment completion (approximately up to 1 year)
Progression-Free Survival (in Part 1b/2) | During the treatment and every 12 weeks after study treatment completion (approximately up to 1 year)
Overall Survival (in Part 1b/2) | During the treatment and every 12 weeks after study treatment completion (approximately up to 1 year)
Time to Response (in Part 1b/2) | During the treatment and every 12 weeks after study treatment completion (approximately up to 1 year)

CONTACTS AND LOCATIONS:
Locations (7):
- Japan (7):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Kobe University Hospital, Kobe, Hyōgo
  - Shizuoka Cancer Center, Nagaizumi-cho, Shizuoka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
  - Osaka International Cancer Institute, Osaka

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated and/or analyzed during the study sponsored by Kyowa Kirin will be available in the Vivli repository, https://vivli.org/ourmember/kyowa-kirin/ as long as conditions of data disclosure specified in the policy section of the Vivli website are satisfied.